CLINICAL TRIAL: NCT03981549
Title: Phase I/II Randomized, Prospective, Double-masked, Sham-controlled Study of Intravitreal Autologous Bone Marrow CD34+ Stem Cell Therapy for Central Retinal Vein Occlusion
Brief Title: Treatment of Central Retinal Vein Occlusion Using Stem Cells Study
Acronym: TRUST
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The Emmes Company, LLC (Industry)
Collaborators: National Eye Institute (NEI) (NIH); University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRUST; 1UG1EY026876-01A1 (NIH); 1UG1EY028517-01 (NIH)
Record Dates: First submitted 2019-06-06; First posted 2019-06-11 (Actual); Results first posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Central Retinal Vein Occlusion
Keywords: Central Retinal Vein Occlusion; Retinal Vein Occlusion; Retinal Diseases; Eye Diseases; CD34+ Stem Cell Therapy; Autologous Bone Marrow Stem Cells; Stem Cells
MeSH Terms: conditions — Retinal Vein Occlusion; Retinal Diseases; Eye Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, examining ophthalmologist, visual acuity examiner, photographers and OCT, perimetry, and ERG technicians will remain masked to study treatment assignment for study duration.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Immediate Cellular Therapy / Deferred Sham Therapy (Active Comparator): At baseline: Bone marrow aspiration followed by intravitreal injection of CD34+ cells.
  At 6 months: Sham bone marrow aspiration and sham intravitreal injection.
  Interventions: Biological: Autologous Bone Marrow CD34+ Stem Cells; Biological: Sham Therapy
- Immediate Sham Therapy / Deferred Cellular Therapy (Sham Comparator): At baseline: Sham bone marrow aspiration followed by sham intravitreal injection.
  At 6 months: Bone marrow aspiration followed by intravitreal injection of CD34+ cells.
  Interventions: Biological: Autologous Bone Marrow CD34+ Stem Cells; Biological: Sham Therapy

INTERVENTIONS:
Biological: Autologous Bone Marrow CD34+ Stem Cells — Single intravitreal injection of autologous bone marrow CD34+ stem cells. The number of cells to be injected per eye will range from 800,000 to 10 million, depending on the yield of the bone marrow aspiration and the isolation procedure.
Biological: Sham Therapy — Sham bone marrow aspiration procedure that penetrates the skin, but does not penetrate the bone followed by sham intravitreal injection without penetration of the eye

SUMMARY:
This study evaluates whether intravitreal autologous CD34+ stem cell therapy is safe, feasible and potentially beneficial in eyes with vision loss from central retinal vein occlusion (CRVO). Half of the participants will receive immediate cellular therapy followed by sham therapy 6 months later, while the other half will receive immediate sham therapy followed by cellular therapy 6 months later. Participants will be followed for a total of 1 year.

DETAILED DESCRIPTION:
The goal of this phase I/II prospective, randomized, sham-controlled, double-masked clinical trial is to determine whether intravitreal autologous CD34+ stem cell therapy is safe, feasible and potentially beneficial in eyes with vision loss from central retinal vein occlusion (CRVO). Retinal Vein Occlusion (RVO) is a leading retinal vascular cause of vision loss in the elderly. CD34+ stem cells in human bone marrow are mobilized into the circulation in response to tissue ischemia for tissue revascularization and repair. Since local delivery of CD34+ stem cells benefits ischemic tissue, intravitreal delivery of CD34+ stem cells may benefit vision and retinal ischemia in eyes with RVO. A pilot clinical trial has shown no major safety or feasibility concerns using intravitreal autologous CD34+ bone marrow stem cells. In this proposed expanded phase I/II study, 20 participants (20 eyes) with persistent vision loss from CRVO will be enrolled and followed for 1 year.

Participants will be randomized 1:1 to immediate cell therapy/deferred sham therapy or immediate sham therapy/deferred cell therapy. At month 6, the cell treated eye will receive sham treatment and the sham treated eye will get cell therapy. The cellular therapy involves bone marrow aspiration, isolation of CD34+ cells from the aspirate under Good Manufacturing Practice (GMP) conditions, and intravitreal injection of isolated CD34+ cells. The sham therapy involves a sham bone marrow aspiration with penetration of the skin but no penetration of the bone and a sham intravitreal injection without penetrating the eye. The participant, examining ophthalmologist, visual acuity examiner, photographers and OCT, perimetry, and electroretinography (ERG) technicians will remain masked to study treatment assignment for study duration. A comprehensive eye examination with ETDRS best-corrected visual acuity, optical coherence tomography (OCT) and OCT angiography (OCTA), autofluorescence, fundus photography, fluorescein angiography, microperimetry, and electroretinography will be performed at baseline and serially. A subset of participants with good fixation on microperimetry and clear media on exam and commercial-grade OCTA and who give consent will have ultra-high resolution cellular retinal imaging using research-grade OCT and OCTA and adaptive optics-OCT at baseline. Participants with high quality images will have repeat imaging at 1 month after stem cell treatment, with at least 2 of the participants randomized to the deferred cellular therapy arm also having imaging 1 month after sham therapy. Post-release flow cytometry characterization will be performed to determine the composition of the CD34+ enriched final product in terms of hematopoietic versus angiogenic stem cells based on cell surface markers (i.e., CD133(+)/CD45(+)/CD34(+) vs CD31(+)/VEGFR-2(+)/CD45(-)/CD34(+)). The long-term objective is to determine whether intravitreal autologous CD34+ cell therapy can minimize, or reverse vision loss associated with retinal ischemia without compromising safety.

ELIGIBILITY:
Study Eye Inclusion/Exclusion Criteria:

Inclusion criteria for the study eye:

* Clinical diagnosis of central retinal vein occlusion (CRVO) confirmed by review of medical records and screening assessment.
* Best Corrected Visual Acuity (BCVA) obtained during the screening period is in the range of 20/40+ to 20/400- (ETDRS letter score in the range of 18 to 73, inclusive).
* Duration of vision loss from CRVO >= 6 months to <=42 months.

Exclusion criteria for the study eye:

* Previous eye treatment with intravitreal or periocular steroids, laser or intraocular surgery within 6 months prior to enrollment (i.e., date ICF signed) or treatment expected to be given during the study period.
* For eyes requiring treatment to prevent recurrent macular edema, on-going intravitreal anti-VEGF treatment is expected to be given at an interval < every 8 weeks during the study period or anti-VEGF therapy was started less than 24 weeks prior to informed consent.
* History of concurrent ocular herpes infection.
* Active non-herpetic eye infection diagnosed within 8 weeks from enrollment (i.e., date Informed Consent Form (ICF) signed).
* Glaucoma requiring treatment with more than 2 medications, laser or intraocular surgery.
* Active uveitis or history of recurrent uveitis or uveitis involving the posterior segment.
* Presence of cataract that is impairing vision.
* Presence of lens or lens implant subluxation.
* History of ocular trauma that is currently impairing vision.
* Any concurrent optic nerve or retinal disease that is visually significant or likely to progress to visual significance during the 1-year study follow-up. The excluded eyes include eyes with AREDS category 2 to 3 age-related macular degeneration (AMD) with foveal involvement of drusen or RPE changes, and any AREDS category 4 AMD eyes. For eyes with ERM, the excluded eyes include eyes with OCT evidence of foveal deformation. For optic nerve disease, eyes with any associated visual field deficit or history of associated CNVM are excluded. For glaucoma eyes, eyes requiring glaucoma laser trabeculectomy or glaucoma surgery to maintain IOP are excluded.
* Active retinal or iris neovascularization.
* Macular edema requiring on-going therapy or where treatment is expected during the study period, with the exception of anti-VEGF treatment given at an interval of 8 weeks or greater.
* Significant media opacity precluding view of the fundus for examination, photography or optical coherence tomography (OCT) including cataract and vitreous haze.
* High myopia (>= 9 diopters)
* Amblyopia
* Other cause contributing to vision loss at screening.
* History of any of the following procedures: corneal transplant, glaucoma surgery, or intraocular silicone oil.

Participant-level Inclusion/Exclusion Criteria:

Participant-level inclusion criteria:

* Age >=18 years
* Female participants of child-bearing potential must not be pregnant or breastfeeding and have a negative urine pregnancy test within 14 days prior to sham injection and/or CD34+ cell injection.
* Females of childbearing potential must have had a hysterectomy, be completely abstinent from intercourse or must agree to practice effective contraception for the duration of the study. Acceptable methods of contraception include hormonal contraception, intrauterine device, barrier methods (diaphragm, condom) with spermicide, or surgical sterilization (tubal ligation).
* Able and willing to sign informed consent.
* Able to keep follow-up appointments for at least 12 months as determined by the investigator.

Participant-level exclusion criteria:

* Concurrent treatment with an investigational drug or device.
* Concurrent use of systemic immunosuppressive therapy or history of use within 3 months prior to enrollment (i.e., date ICF signed).
* Concurrent use of anticoagulation therapy except for aspirin without an acceptable safe stopping plan for study treatments.
* Known history of coagulopathy or other hematologic abnormality that may put participant at risk for bleeding or infection or raise concerns about quality or quantity of CD34+ cells isolated.
* History of allergy to fluorescein dye.
* Participant who has had a prior or concomitant malignancy with the exception of the following: 1) adequately treated basal or squamous cell carcinoma of the skin, or 2) any other malignancy from which the patient has remained disease free for more than five years.
* Current active systemic infection as evidenced by fever greater than 100.4 or any evidence of systemic infection as determined by the study physician.
* Any diagnosis of active infection or vaccination within 8 weeks of study treatment.
* Diabetes mellitus with known systemic complications by self-report or physician-determined by medical history or examination.
* History of prior radiotherapy to head/neck area.
* Poorly controlled hypertension with systolic > 180 or diastolic > 95.
* Serious medical or psychiatric condition that, in the opinion of the Investigator, would make study participation hazardous to the participant or compromise study findings or would prevent the participant from completing the study.
* Any physical characteristic that precludes ability to perform study diagnostic testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-11-07 (Actual); Study Completion 2023-11-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna S Park, MD, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Department of Ophthalmology & Vision Science, University of California Davis Eye Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: Yes
TRUST will follow specific plans for sharing of research data under the guidance of NIH's 2003 Data Sharing Policy. After analysis, the final data set can be provided after appropriate procedures are implemented to preserve the anonymity of the records, specifically where protected health information (PHI) is required. Upon request, anonymized data will be shared under confidentiality agreements with researchers interested in the project.
Supporting Information: Study Protocol, SAP
Time Frame: Time Frame will be determined.
Access Criteria: Confidentiality agreements will be required before anonymized data will be shared.

REFERENCES:
- [Background] Park SS, Bauer G, Abedi M, Pontow S, Panorgias A, Jonnal R, Zawadzki RJ, Werner JS, Nolta J. Intravitreal autologous bone marrow CD34+ cell therapy for ischemic and degenerative retinal disorders: preliminary phase 1 clinical trial findings. Invest Ophthalmol Vis Sci. 2014 Dec 9;56(1):81-9. doi: 10.1167/iovs.14-15415. PMID 25491299
- [Background] Park SS, Bauer G, Fury B, Abedi M, Perotti N, Colead-Bergum D, Nolta JA. Phase I Study of Intravitreal Injection of Autologous CD34+ Stem Cells from Bone Marrow in Eyes with Vision Loss from Retinitis Pigmentosa. Ophthalmol Sci. 2024 Jul 31;5(1):100589. doi: 10.1016/j.xops.2024.100589. eCollection 2025 Jan-Feb. PMID 39328826
- [Derived] Romano F, Lamanna F, Gabrielle PH, Teo KYC, Battaglia Parodi M, Iacono P, Fraser-Bell S, Cornish EE, Nassisi M, Viola F, Agarwal A, Samanta A, Chhablani J, Staurenghi G, Invernizzi A. Update on Retinal Vein Occlusion. Asia Pac J Ophthalmol (Phila). 2023 Mar-Apr 01;12(2):196-210. doi: 10.1097/APO.0000000000000598. Epub 2023 Feb 14. PMID 36912792

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Cellular Therapy / Deferred Sham Therapy: At baseline: Bone marrow aspiration followed by intravitreal injection of CD34+ cells.
  At 6 months: Sham bone marrow aspiration and sham intravitreal injection.
  Autologous Bone Marrow CD34+ Stem Cells: Single intravitreal injection of autologous bone marrow CD34+ stem cells. The number of cells to be injected per eye will range from 800,000 to 10 million, depending on the yield of the bone marrow aspiration and the isolation procedure.
  Sham Therapy: Sham bone marrow aspiration procedure that penetrates the skin, but does not penetrate the bone followed by sham intravitreal injection without penetration of the eye
- Immediate Sham Therapy / Deferred Cellular Therapy: At baseline: Sham bone marrow aspiration followed by sham intravitreal injection.
  At 6 months: Bone marrow aspiration followed by intravitreal injection of CD34+ cells.
  Autologous Bone Marrow CD34+ Stem Cells: Single intravitreal injection of autologous bone marrow CD34+ stem cells. The number of cells to be injected per eye will range from 800,000 to 10 million, depending on the yield of the bone marrow aspiration and the isolation procedure.
  Sham Therapy: Sham bone marrow aspiration procedure that penetrates the skin, but does not penetrate the bone followed by sham intravitreal injection without penetration of the eye
Period: Overall Study
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy | Total
Number analyzed (Participants) | 7 | 9 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (12.59) | 62.7 (12.62) | 64.9 (12.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 4 | 7 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 8 | 15
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 7 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Ocular and Systemic Adverse Events
Description: The primary safety outcome will be assessed at month 6. Adverse events (AE) that occur during the first 6 months of the trial will be broken down by whether the AE occurred following the sham or cellular treatment to assess differences in the adverse event experience between the cellular and sham therapies.
Time Frame: Months 0 to 6
Population: Number of participants randomized
Measure: Number; unit: participants
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
participants
  Altered visual depth perception in study eye | 1 | 0
  Chalazion in study eye | 0 | 1
  Cystoid macular oedema in study eye | 0 | 1
  Dermatochalasis in study eye | 0 | 1
  Dry eye in study eye | 2 | 4
  Eye irritation in study eye | 5 | 4
  Eye pain in study eye | 4 | 2
  Eye puritis in study eye | 1 | 1
  Foreign body sensation in study eye | 2 | 3
  Meibomian gland dysfuntion in study eye | 1 | 1
  Ocular hyperaemia in study eye | 3 | 3
  Periorbital irritation in study eye | 0 | 1
  Photopsia in study eye | 0 | 1
  Presbyopia in study eye | 1 | 0
  Swelling of eyelid in study eye | 1 | 0
  Vision blurred in study eye | 1 | 1
  Visual acuity reduced in study eye | 0 | 1
  Visual impairment in study eye | 2 | 0
  Vitreous degeneration in study eye | 1 | 0
  Vitreous detachment in study eye | 1 | 0
  Vitreous floaters in study eye | 6 | 0
  Cystoid macular oedema in fellow eye | 0 | 1
  Visual impairment in fellow eye | 1 | 1
  Vitreous floaters in fellow eye | 1 | 1
  Abdominal pain upper | 0 | 1
  Acarodermatitis | 0 | 1
  Anaemia | 0 | 1
  Appendicitis | 0 | 1
  Arthralgia | 1 | 0
  Arthropod bite | 1 | 0
  Back pain | 1 | 1
  Basal cell carcinoma | 1 | 0
  Cholelithiasis | 1 | 0
  Chronic kidney disease | 1 | 0
  Dizziness | 1 | 0
  Epicondylitis | 0 | 1
  Fall | 0 | 3
  Foot deformity | 0 | 1
  Heat exhaustion | 0 | 1
  Hypertension | 2 | 0
  Immunisation reaction | 1 | 3
  Migraine | 0 | 1
  Neuralgia | 1 | 0
  Osteoarthritis | 1 | 0
  Pain in extremity | 1 | 0
  Palpitations | 1 | 0
  Procedural pain | 0 | 1
  Rash | 0 | 1
  Rectal haemorrhage | 0 | 1
  Rib fracture | 0 | 1
  Sciatica | 0 | 1
  Soft tissue mass | 1 | 0
  Squamous cell carcinoma of skin | 1 | 0
  Upper respiratory tract infection | 1 | 1
  White blood cell count decreased | 1 | 0

2. Primary Outcome: Feasibility of the Stem Cell Therapy
Description: Number of CD34+ cells isolated from the bone marrow aspirate and number of cells injected into the eye
Time Frame: Day 0 and Day 182
Population: All participants with successful bone marrow aspiration
Measure: Mean (Standard Deviation); unit: Number of cells in millions
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
Number of cells in millions
  Number of CD34+ cells isolated from the bone marrow aspirate (pre-release) | 5.4 (2.20) | 5.9 (4.65)
  Number of CD34+ cells injected into the eye (pre-release) | 3.8 (1.69) | 4.6 (4.14)

3. Secondary Outcome: Change in Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity Letter Score
Description: Mean change from baseline of visual acuity letter score at Month 6. The measure is calculated by subtracting the baseline visual acuity letter score from the month 6 visual acuity letter score. The participant is refracted for best corrected vision, and then reads single letters from the ETDRS charts using a visual acuity light box at a 4 meter distance (or 1 meter for participants with sufficiently reduced vision) according to a specific algorithm. A letter score is provided that ranges from 0 (unable to read any letters) to 100. A visual acuity letter score of 85 corresponds to a visual acuity of 20/20 as a Snellen equivalent. Higher is better.
Time Frame: Months 0 to 6
Population: All participants with visual acuity letter score recorded at Month 6
Measure: Mean (Standard Deviation); unit: Letters read
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
Letters read | 1.7 (3.82) | 2.1 (10.98)

4. Secondary Outcome: Change in % Reduced Sensitivity
Description: Mean change from baseline of % reduced sensitivity at Month 6 as measured by microperimetry (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with reduced sensitivity recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent reduced
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent reduced | 0.8 (14.00) | -11.4 (16.81)

5. Secondary Outcome: Change in Average Threshold
Description: Mean change from baseline of average threshold (dB) at Month 6 as measured by microperimetry (increase is better)
Time Frame: Months 0 to 6
Population: All participants with average threshold recorded at Month 6
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
dB | -1.2 (2.99) | 0.0 (3.83)

6. Secondary Outcome: Change in Percent Normal Amplitude for ERG+OP (Oscillatory Potential) A-wave Under Scotopic Conditions
Description: Mean change from baseline of percent of normal amplitude for ERG+OP a-wave under scotopic conditions at Month 6 as measured by Full-field ERG (increase is better)
Time Frame: Months 0 to 6
Population: All participants with normal amplitude for ERG+OP a-wave under scotopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal amplitude
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 8
percent normal amplitude | -7.7 (36.84) | 18.6 (18.15)

7. Secondary Outcome: Change in Percent Normal Amplitude for ERG+OP B-wave Under Scotopic Conditions
Description: Mean change from baseline of percent of normal amplitude for ERG+OP b-wave under scotopic conditions at Month 6 as measured by Full-field ERG (increase is better)
Time Frame: Months 0 to 6
Population: All participants with normal amplitude for ERG+OP b-wave under scotopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal amplitude
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 8
percent normal amplitude | -8.4 (48.94) | 11.6 (22.50)

8. Secondary Outcome: Change in Percent Normal Latency of ERG+OP A-wave Under Scotopic Conditions
Description: Mean change from baseline of percent normal latency of ERG+OP a-wave under scotopic conditions at Month 6 as measured by Full-field ERG (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with normal latency for a-wave under scotopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal latency
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 8
percent normal latency | 1.3 (21.59) | -9.0 (8.33)

9. Secondary Outcome: Change in Percent Normal Latency of ERG+OP B-wave Under Scotopic Conditions
Description: Mean change from baseline of percent normal latency of ERG+OP b-wave under scotopic conditions at Month 6 as measured by Full-field ERG (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with normal latency of ERG+OP b-wave under scotopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal latency
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 8
percent normal latency | 12.7 (42.38) | -1.2 (24.95)

10. Secondary Outcome: Change in Percent Normal Amplitude for A-wave Under Photopic Conditions
Description: Mean change from baseline of percent normal amplitude for a-wave under photopic conditions at Month 6 as measured by Full-field ERG (increase is better)
Time Frame: Months 0 to 6
Population: All participants with normal amplitude for a-wave under photopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal amplitude
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent normal amplitude | 6.2 (35.84) | 26.8 (79.01)

11. Secondary Outcome: Change in Percent Normal Amplitude for B-wave Under Photopic Conditions
Description: Mean change from baseline of percent normal amplitude for b-wave under photopic conditions at Month 6 as measured by Full-field ERG (increase is better)
Time Frame: Months 0 to 6
Population: All participants with normal amplitude for b-wave under photopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal amplitude
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent normal amplitude | -2.5 (21.83) | -6.0 (22.83)

12. Secondary Outcome: Change in Percent Normal Latency for A-wave Under Photopic Conditions
Description: Mean change from baseline of percent normal latency for a-wave under photopic conditions at Month 6 as measured by Full-field ERG (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with normal latency for a-wave under photopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal latency
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent normal latency | -3.5 (20.19) | -0.0 (13.08)

13. Secondary Outcome: Change in Percent Normal Latency for B-wave Under Photopic Conditions
Description: Mean change from baseline of percent normal latency for b-wave under photopic conditions at Month 6 as measured by Full-field ERG (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with normal latency for b-wave under photopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal latency
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent normal latency | -0.1 (10.26) | -4.7 (7.59)

14. Secondary Outcome: Change in Percent Normal Flicker Amplitude
Description: Mean change from baseline in percent normal flicker amplitude at Month 6 as measured by Full-field ERG (increase is better)
Time Frame: Months 0 to 6
Population: All participants with normal flicker amplitude recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal flicker amplitude
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent normal flicker amplitude | -10.8 (14.10) | 2.2 (15.08)

15. Secondary Outcome: Change in Flicker Latency Trough
Description: Mean change from baseline of latency trough at Month 6 as measured by Full-field ERG (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with latency trough recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent latency trough
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent latency trough | -4.2 (8.92) | -0.3 (8.12)

16. Secondary Outcome: Change in Percent Normal Amplitude for A-wave Under Scotopic Conditions
Description: Mean change from baseline of percent normal amplitude for a-wave under scotopic conditions at Month 6 as measured by Full-field ERG (increase is better)
Time Frame: Months 0 to 6
Population: All participants with normal amplitude for a-wave under scotopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal amplitude
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent normal amplitude | 8.2 (42.65) | 3.8 (48.29)

17. Secondary Outcome: Change in Percent Normal Latency of A-wave Under Scotopic Conditions
Description: Mean change from baseline of percent normal latency of a-wave under scotopic conditions at Month 6 as measured by Full-field ERG (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with normal latency of a-wave under scotopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal latency
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent normal latency | 12.4 (56.19) | -14.7 (24.81)

18. Secondary Outcome: Change in Percent Normal Amplitude for B-wave Under Scotopic Conditions
Description: Mean change from baseline of percent normal amplitude for b-wave under scotopic conditions at Month 6 as measured by Full-field ERG (increase is better)
Time Frame: Months 0 to 6
Population: All participants with normal amplitude for b-wave under scotopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal amplitude
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent normal amplitude | -1.7 (35.75) | 19.2 (34.67)

19. Secondary Outcome: Change in Percent Normal Latency for B-wave Under Scotopic Conditions
Description: Mean change from baseline of percent normal latency for b-wave under scotopic conditions at Month 6 as measured by Full-field ERG (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with normal latency for b-wave under scotopic conditions recorded at Month 6
Measure: Mean (Standard Deviation); unit: percent normal latency
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
percent normal latency | -4.9 (12.32) | -5.7 (14.47)

20. Secondary Outcome: Foveal Avascular Zone Integrity
Description: Number of study eyes in each of the following categories as it relates to the integrity of the foveal avascular zone: Intact, Questionable, Disrupted (<900 microns), Disrupted (900-1800 microns), Disrupted (>1800 microns), and Cannot grade. Measured at Month 6 by fluorescein angiogram
Time Frame: 6 months
Population: All participants with integrity of the foveal avascular zone recorded at Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 9
Participants
  Foveal Avascular Zone Integrity at Baseline: Intact | 0 | 1
  Foveal Avascular Zone Integrity at Baseline: Questionable | 2 | 2
  Foveal Avascular Zone Integrity at Baseline: Disrupted (<900 microns) | 1 | 2
  Foveal Avascular Zone Integrity at Baseline: Disrupted (900-1800 microns) | 1 | 4
  Foveal Avascular Zone Integrity at Baseline: Disrupted (>1800 microns) | 3 | 0
  Foveal Avascular Zone Integrity at Baseline: Cannot grade | 0 | 0
  Foveal Avascular Zone Integrity at Month 6: Intact | 0 | 2
  Foveal Avascular Zone Integrity at Month 6: Questionable | 2 | 0
  Foveal Avascular Zone Integrity at Month 6: Disrupted (<900 microns) | 2 | 2
  Foveal Avascular Zone Integrity at Month 6: Disrupted (900-1800 microns) | 2 | 4
  Foveal Avascular Zone Integrity at Month 6: Disrupted (>1800 microns) | 1 | 0
  Foveal Avascular Zone Integrity at Month 6: Cannot grade | 0 | 1

21. Secondary Outcome: Change in Area of Non-perfusion Within ETDRS Grid
Description: Mean change from baseline of area of non-perfusion within ETDRS grid at Month 6 as measured by fluorescein angiogram (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with area of non-perfusion within ETDRS grid recorded at Month 6
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 7 | 8
mm^2 | 1.4 (2.54) | -3.3 (6.32)

22. Secondary Outcome: Change in Area of Non-perfusion Within Networc Grid
Description: Mean change from baseline of area of non-perfusion within Networc grid at Month 6 as measured by fluorescein angiogram (decrease is better)
Time Frame: Months 0 to 6
Population: All participants with area of non-perfusion within Networc grid recorded at Month 6
Measure: Mean (Standard Deviation); unit: mm^2
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy | Immediate Sham Therapy / Deferred Cellular Therapy
Number analyzed (Participants) | 6 | 5
mm^2 | 0.2 (152.70) | 28.0 (53.61)

ADVERSE EVENTS:
Time Frame: Baseline to Month 12
Description: The safety of the intravitreal injection of autologous CD34+ cells was assessed through regular eye examinations during the 12 month follow-up period. Adverse events (AEs) including new or worsening ocular conditions that occured from the time the participant signed informed consent until the final study visit were recorded, regardless of suspected cause. An AE and/or serious adverse event form was completed and the information was entered into the study electronic data capture system.
Groups:
- Immediate Cellular Therapy / Deferred Sham Therapy: Months 0-6: Data for Month 0 through Month 6. Treatment arms defined as follows.
  At baseline: Bone marrow aspiration followed by intravitreal injection of CD34+ cells.
  At 6 months: Sham bone marrow aspiration and sham intravitreal injection.
  Autologous Bone Marrow CD34+ Stem Cells: Single intravitreal injection of autologous bone marrow CD34+ stem cells. The number of cells to be injected per eye will range from 800,000 to 10 million, depending on the yield of the bone marrow aspiration and the isolation procedure.
  Sham Therapy: Sham bone marrow aspiration procedure that penetrates the skin, but does not penetrate the bone followed by sham intravitreal injection without penetration of the eye
- Immediate Sham Therapy / Deferred Cellular Therapy: Months 0-6: Data for Month 0 through Month 6. Treatment arms defined as follows.
  At baseline: Sham bone marrow aspiration followed by sham intravitreal injection.
  At 6 months: Bone marrow aspiration followed by intravitreal injection of CD34+ cells.
  Autologous Bone Marrow CD34+ Stem Cells: Single intravitreal injection of autologous bone marrow CD34+ stem cells. The number of cells to be injected per eye will range from 800,000 to 10 million, depending on the yield of the bone marrow aspiration and the isolation procedure.
  Sham Therapy: Sham bone marrow aspiration procedure that penetrates the skin, but does not penetrate the bone followed by sham intravitreal injection without penetration of the eye
- Immediate Cellular Therapy / Deferred Sham Therapy: Months 6-12: Data for Month 6 through Month 12. Treatment arms defined as follows.
  At baseline: Bone marrow aspiration followed by intravitreal injection of CD34+ cells.
  At 6 months: Sham bone marrow aspiration and sham intravitreal injection.
  Autologous Bone Marrow CD34+ Stem Cells: Single intravitreal injection of autologous bone marrow CD34+ stem cells. The number of cells to be injected per eye will range from 800,000 to 10 million, depending on the yield of the bone marrow aspiration and the isolation procedure.
  Sham Therapy: Sham bone marrow aspiration procedure that penetrates the skin, but does not penetrate the bone followed by sham intravitreal injection without penetration of the eye
- Immediate Sham Therapy / Deferred Cellular Therapy: Months 6-12: Data for Month 6 through Month 12. Treatment arms defined as follows.
  At baseline: Sham bone marrow aspiration followed by sham intravitreal injection.
  At 6 months: Bone marrow aspiration followed by intravitreal injection of CD34+ cells.
  Autologous Bone Marrow CD34+ Stem Cells: Single intravitreal injection of autologous bone marrow CD34+ stem cells. The number of cells to be injected per eye will range from 800,000 to 10 million, depending on the yield of the bone marrow aspiration and the isolation procedure.
  Sham Therapy: Sham bone marrow aspiration procedure that penetrates the skin, but does not penetrate the bone followed by sham intravitreal injection without penetration of the eye
Arm/Group | Immediate Cellular Therapy / Deferred Sham Therapy: Months 0-6 | Immediate Sham Therapy / Deferred Cellular Therapy: Months 0-6 | Immediate Cellular Therapy / Deferred Sham Therapy: Months 6-12 | Immediate Sham Therapy / Deferred Cellular Therapy: Months 6-12
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/9 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 1/9 | 1/7 | 0/9
Other Adverse Events (participants affected / at risk) | 7/7 | 9/9 | 7/7 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Cellular Therapy / Deferred Sham Therapy: Months 0-6 (N=7) | Immediate Sham Therapy / Deferred Cellular Therapy: Months 0-6 (N=9) | Immediate Cellular Therapy / Deferred Sham Therapy: Months 6-12 (N=7) | Immediate Sham Therapy / Deferred Cellular Therapy: Months 6-12 (N=9)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Iris Neovascularization (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immediate Cellular Therapy / Deferred Sham Therapy: Months 0-6 (N=7) | Immediate Sham Therapy / Deferred Cellular Therapy: Months 0-6 (N=9) | Immediate Cellular Therapy / Deferred Sham Therapy: Months 6-12 (N=7) | Immediate Sham Therapy / Deferred Cellular Therapy: Months 6-12 (N=9)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Altered visual depth perception (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract cortical (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cystoid macular oedema (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Dermatochalasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 2 (2) | 4 (4) | 0 (0) | 2 (3)
Eye irritation (Eye disorders) | 5 (5) | 4 (5) | 3 (3) | 4 (6)
Eye pain (Eye disorders) | 4 (4) | 2 (2) | 3 (3) | 4 (4)
Eye pruritus (Eye disorders) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 2 (2) | 3 (3) | 4 (4) | 4 (6)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meibomian gland dysfunction (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 3 (3) | 3 (4) | 4 (4) | 5 (5)
Periorbital irritation (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presbyopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Retinal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling of eyelid (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (3) | 1 (1) | 2 (2) | 1 (1)
Visual acuity reduced (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Visual impairment (Eye disorders) | 3 (5) | 1 (1) | 3 (3) | 2 (3)
Vitreous degeneration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vitreous floaters (Eye disorders) | 6 (10) | 1 (1) | 0 (0) | 9 (9)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epicondylitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Heat exhaustion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1) | 3 (4)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Foot deformity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Soft tissue mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Panic attack (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth extraction (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/49/NCT03981549/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-02): https://cdn.clinicaltrials.gov/large-docs/49/NCT03981549/SAP_001.pdf